CLINICAL TRIAL: NCT03091140
Title: Alterations in Muscle's Functional Characteristics After Parathyroid Surgery for Primary Hyperparathyroidism.
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Assistant Professor of Surgery, Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Other Study IDs: 29th SesTop/31stCon/21.12.2016
Record Dates: First submitted 2017-03-03; First posted 2017-03-27 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hyperparathyroidism, Primary; Parathyroidectomy
Keywords: Parathyroidectomy; Muscular Functional Characteristics; Parathyroid Glands
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: patients with primary hyperparathyroidism, undergoing parathyroidectomy, as a therapeutic intervention
- Group B: patients with primary hyperparathyroidism, not undergoing parathyroidectomy and receiving conservative treatment. This group will be considered as control group.
- Group C: patients undergoing thyroid surgery due to nontoxic multinodular goiter or solitary nontoxic thyroid adenoma. This group will be considered as control group.
- Group D: healthy subjects. This group will be considered as control group.

SUMMARY:
Protocol title: Alterations in functional characteristics of the muscle tissue following surgery for primary hyperparathyroidism.

Purpose: To detect any changes in functional characteristics of muscles in patients who undergo surgery for primary hyperparathyroidism compared to patients with primary hyperparathyroidism and conservative treatment, patients undergoing thyroid surgery and healthy subjects.

Design: Prospective, multi-center observational study Patient Population: Male or female subjects 18 years of age or older scheduled for parathyroidectomy No. of Subjects: 50 patients undergoing parathyroidectomy, 50 patients undergoing conservative follow up, 50 patients undergoing thyroid surgery due to nontoxic multinodular goiter or solitary nontoxic thyroid adenoma and 50 healthy control subjects, estimated up to 12 months to enroll.

Duration of Treatment: During the operation Duration of Follow-up: Follow-up will be performed daily during hospitalization and at 3, 6 and 12 months after the procedure Endpoints: To evaluate the changes in functional characteristics of all the type of muscles which occur after parathyroidectomy for primary hyperparathyroidism.

DETAILED DESCRIPTION:
1.0 INTRODUCTION The association between parathyroidectomy and cardiovascular status improvement is still inconclusive. There is evidence to suggest that primary hyperparathyroidism (PHPT) is associated with hypertension, whereas few studies show that hypertension does not reverse after surgical care. Moreover, left ventricular hypertrophy (LVH) is considered to be linearly associated with parathyroid hormone (PTH) and independent of hypertension. In addition, inflammatory changes in the cardiovascular system, which are expected to occur after parathyroidectomy, can be evaluated by assessing the levels of inflammation biomarkers, such as high-sensitivity C reactive protein (hs-CRP), increased levels of which are associated with high cardiovascular event rate. The investigators will evaluate cardiovascular system before and after parathyroidectomy by appraising the levels of hs-CRP, measuring Left Ventricular Mass Index (LVMI) and monitoring patients' blood pressure (BP) for 24 hours.

Primary hyperparathyroidism (PHPT) has also been associated with neuromuscular abnormalities. The typical symptoms are proximal muscle weakness and muscle atrophy, especially of type II fibers. Other symptoms are generalized fatigue, reduced well-being, hyperreflexia, abnormal gait and tongue fasciculations. Although, nowadays, most of the symptoms with which patients are presented are mild or completely absent probably because PHPT is detected at a preclinical stage. On the other hand, many "asymptomatic" patients preoperatively, report subjective amelioration after the surgery, with respect to muscle strength and function. The investigators will conduct clinical examination, focusing on neuromuscular status, assess motor nerve conduction velocity, using electroneurography (ENG) and muscle strength, using isokinetic dynamometers. Moreover, the investigators will evaluate neuromuscular junction with the help of electrodiagnostic techniques, such as electromyography (EMG). Finally, due to the fact that stapedius muscle is the smallest skeletal muscle in the human body, the investigators tend to measure stapedius reflex in order to test the hypothesis that there is association between acoustic reflex improvement and parathyroidectomy for PHPT.

2.0 OBJECTIVES To detect and compare the changes in functional characteristics of muscles, which occur in patients who undergo surgery for primary hyperparathyroidism compared to patients with primary hyperparathyroidism and conservative treatment, patients undergoing thyroid surgery and healthy subjects.

3.0 DESIGN AND STUDY POPULATION The study is designed as a prospective, multi-center, observational study. Any patient that has indication for a parathyroidectomy, as a therapeutic intervention, due to primary hyperparathyroidism will be considered eligible.

3.1 Duration of the study The study will be conducted until all subjects of each category are included. It is estimated that it will take up to 12 months to enroll the patients and an additional 12 months to obtain the follow-up information

4.0 STUDY PROCEDURE

4.1 Pre-Surgery

Procedures performed such as routine hospital examinations, antibiotic prophylactic treatment, anticoagulant treatment and diet will be according to the standard management protocol and will be recorded for the study. The following pre-surgery information will be recorded:

1. Demographic information including: name, age, gender, ethnicity
2. Height, weight, BMI and American Society of Anesthesiologists physical status classification system (I-VI)
3. Behavioral history (Smoking, alcohol or drug use)
4. Blood Pressure and Ultra Sound measurement of Left Ventricular Mass Index (LVMI)
5. Neurological clinical examination
6. Hearing and stapedius reflex assessment
7. Electromyography and electroneurography
8. Muscle strength status
9. Preoperative labs [white blood cells (WBC), hematocrit (Ht), hemoglobin (Hgb), serum calcium (Ca2+), free triiodothyronine (fT3), free thyroxine (fT4), thyroid-stimulating hormone (TSH), PTH, vitamin D (VitD), creatine phosphokinase (CPK), lactate dehydrogenase (LDH), hs-CRP]
10. Diagnosis including clinical observations and previous imaging results
11. Pre-operative characteristics of the adenoma
12. Medications
13. Questionnaire assessing subjects' physical activity
14. Current and past history of surgical and medical comorbidities

4.2 Intra-operative

The surgeon will perform the preplanned operation. The following intraoperative variables will be recorded for all patients:

1. Surgery date
2. Duration of surgery
3. Operation performed
4. Procedure related comments
5. Intraoperative frozen section
6. Quick intraoperative parathyroid assay (intact PTH intra-operative values)

4.3 Pathology data form

The following pathology data will be recorded for all patients:

1. Post-operative diagnosis including pathology report
2. Weight of the adenoma
3. Dimensions of the adenoma

4.4 Postoperative follow-up

Follow-up evaluation will be performed during hospitalization, at the 3rd, 6th and 12th month. The following information will be recorded:

1. Postoperative labs (WBC, Ht, Hgb, Ca2+, fT3, fT4, TSH, PTH, VitD, CPK, LDH, Hs- CRP)
2. Blood Pressure and Ultra Sound measurement of Left Ventricular Mass Index (LVMI)
3. Neurological clinical examination
4. Hearing and stapedius reflex assessment
5. Electromyography and electroneurography
6. Muscle strength status
7. Questionnaire assessing subjects' physical activity
8. Comments

5.0 COMPLICATIONS AND ADVERSE EVENTS

The investigator is required to notify the Ethics Committee of any serious adverse events, according to local regulations and requirements. Serious Adverse Events include:

1. Death regardless of cause
2. Any-life-threatening event
3. Any hospitalization or prolongation of existing hospitalization
4. Any event that results in persistent or significant disability or incapacity to the patient.

6.0 STATISTICAL ANALYSIS The objective of this study is to detect and compare the changes in functional characteristics of muscles, which occur in patients who undergo surgery for primary hyperparathyroidism comparing with patients who do not, patients undergoing thyroid surgery and healthy subjects. All the subject will be matched in race, gender and age.

Four groups will be formed:

1. Group A, which includes patients with PHPT, undergoing parathyroidectomy, as a therapeutic intervention.
2. Group B, which includes patients with PHPT, not undergoing parathyroidectomy and receiving conservative treatment. This group will be considered as control group.
3. Group C, which includes patients undergoing thyroid surgery due to nontoxic multinodular goiter or solitary nontoxic thyroid adenoma. This group will be considered as control group.
4. Group D, which includes healthy subjects. This group will be considered as control group.

In order to efficiently evaluate the contribution of parathyroidectomy for PHPT in the functional alterations occurring after it, the investigators will search for significant statistical differences in pre- and postoperative alterations in muscles' functional characteristics in Group A, using repeated measure ANOVA for continuous variables and Cochran's Q test for categorical data.

Furthermore, differences in functional characteristics of muscles between the four groups will be explored using ANOVA for continuous data and Fischer's Exact Test for categorical data. Baseline characteristics will be summarized using appropriate descriptive statistics. Statistical significance will be set at 0.05.

Since the study does not have pre-specified hypotheses all statistical analyses are exploratory and interpretation of results should be within this context.

7.0 DATA MONITORING PLAN The investigators are going to monitor all data accrual. Furthermore, the investigators will review the progress of the clinical trial including safety data and ensure as possible that it is conducted, recorded and reported in accordance with the protocol, good clinical practice and the applicable regulatory requirements.

8.0 DATA CONFIDENTIALITY Each patient will be identified by his/her initials and a unique patient identification number. Source data will be stored with source documents. Only personnel responsible for collecting data and transcribing it into the case report forms will have access to the data. Records will remain on site in secure areas.

9.0 FUNDING No additional funding for the execution of the present protocol is necessary. The investigators are willing to execute the present study without any additional reimbursement.

10.0 ETHICS Prior to study institution review board (IRB) approval should be obtained. Any changes in the study protocol, informed consent forms, or investigator must be re-approved by the IRB. All patients enrolled in the study will provide their consent prior to entering the study. An informed consent form shall be signed and dated by the patient. The investigator will retain the forms as part of the study records.

This study will be executed in accordance with the Declaration of Helsinki, in agreement with the guidelines for conducting a clinical investigation in accordance with the principles of ICH (International Conference on Harmonization) GCP (Good Clinical Practice) outlined in the E6 document. By signing the present protocol, participants in the study commit themselves to carry it out in accordance with local legal requirements.

11.0 INFORMED CONSENT All eligible patients should have the capacity to provide an informed consent. The above described inclusion and exclusion criteria were designed to ensure the entry of the appropriate population of patients to this study and will be approved by the local IRB. Screening for these criteria will be conducted by the coordinator. Eligible patients will be educated about the research proposal by a study investigator. To determine whether the patient has understood the issues, he/she will be asked to describe what the research entails and whether they have any questions. All questions will be addressed prior to enrollment. The patient can refuse participation in the study at any time. A written informed consent form will be generated. For each patient, a case report form (CRF) will be completed, providing general medical information and history.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient scheduled for a non-emergency operation
3. Patients diagnosed with PHPT:

   i) one or more samples of total serum calcium above the upper limit of normal value for the laboratory (hypercalcemia) ii) serum albumin within the normal range iii) hypercalcemia with normal or elevated PTH levels iv) serum 25(OH) vitamin D more than 20 ng/ml (50nmol/lt)
4. Patient eligible for parathyroid surgery: PHPT with one or more of the following i) age less than 50 years ii) serum calcium level more than 1mg/dl above the upper limit of normal iii) T score of less than -2.5 at any site, or non traumatic osteoporotic fracture by history or VFA (Vertebral Fracture Assessment) iv) history of renal colic or evidence of lithiasis/calcinosis by x-Ray or ultrasound v) creatinine clearance of less than 60ml/min vi) hypercalciuria (more than 400mg/ day)
5. Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion Criteria:

1. Patient is participating in another clinical trial which may affect this study's outcomes
2. Patient with recurrent hyperparathyroidism
3. Previous operation at the thyroid and parathyroid glands or neck irradiation
4. Noneuthyroid condition
5. Primary hyperparathyroidism due to hyperplasia or multiple adenomas
6. Secondary hyperparathyroidism
7. Primary or secondary hypoparathyroidism
8. Diabetes mellitus
9. Chronic renal failure
10. Systemic diseases (e.g. infections, neoplasms)
11. Hypoalbuminemia
12. Use of drugs that influences calcium metabolism (Vitamin D analogues, oral calcium supplements, bisphosphonates, teriparatide, thiazide diuretics, aromatase inhibitors)
13. Known neuromuscular disorders due to other causes
14. Factors affecting acoustic reflex:

    i) Conductive or sensorineural hearing loss (hearing threshold better than 80dBs (decibells) in every testing frequency) ii) Otosclerosis iii) Middle ear dysfunction (acute or chronic inflammation) iv) Facial nerve dysfunction v) Retrocochlear damage (acoustic neurinoma, vestibular Schwannoma) vi) Impaired stapedius muscle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is designed as a multi-center, observational, cohort study. Any patient that has indication for a parathyroidectomy due to primary hyperparathyroidism will be considered eligible.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring stapedius reflex. | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  Due to the fact that stapedius muscle is the smallest skeletal muscle in the human body, the investigators tend to measure stapedius reflex in order to test the hypothesis that there is association between acoustic reflex improvement and parathyroidectomy for PHPT.
Measuring Left Ventricular Mass Index | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  Cardiovascular system will be evaluated by measuring Left Ventricular Mass Index (LVMI)
Assessing muscle strength. | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  The investigators will assess muscle strength using isokinetic dynamometers

SECONDARY OUTCOMES:
Measuring the levels of hs-CRP | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  Concerning evaluation of cardiovascular system, the investigators will also appraise the levels of hs-CRP
Monitoring patients' blood pressure for 24 hours. | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  Concerning evaluation of cardiovascular system, the investigators will also monitor patients' blood pressure for 24 hours.
Neurological assessment | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  The investigators will conduct neurological clinical examination and assess motor nerve conduction velocity, using electroneurography and neuromuscular junction, using electromyography
Assessing quality of life | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  Pasiekas' questionnaire will be used to assess participant's quality of life.
Assessing physical activity | It will be assessed before surgery and at 3, 6 and 12 months after parathyroidectomy
  International Physical Activity questionnaire will be used to assess participant's physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Theodossis Papavramidis, Ass. Professor, Study Director — 1st Propedeutic Department of Surgery, AHEPA University General Hospital, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University General Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farahnak P, Ring M, Caidahl K, Farnebo LO, Eriksson MJ, Nilsson IL. Cardiac function in mild primary hyperparathyroidism and the outcome after parathyroidectomy. Eur J Endocrinol. 2010 Sep;163(3):461-7. doi: 10.1530/EJE-10-0201. Epub 2010 Jun 18. PMID 20562163
- [Background] Walker MD, Rundek T, Homma S, DiTullio M, Iwata S, Lee JA, Choi J, Liu R, Zhang C, McMahon DJ, Sacco RL, Silverberg SJ. Effect of parathyroidectomy on subclinical cardiovascular disease in mild primary hyperparathyroidism. Eur J Endocrinol. 2012 Aug;167(2):277-85. doi: 10.1530/EJE-12-0124. Epub 2012 Jun 1. PMID 22660025
- [Background] Piovesan A, Molineri N, Casasso F, Emmolo I, Ugliengo G, Cesario F, Borretta G. Left ventricular hypertrophy in primary hyperparathyroidism. Effects of successful parathyroidectomy. Clin Endocrinol (Oxf). 1999 Mar;50(3):321-8. doi: 10.1046/j.1365-2265.1999.00651.x. PMID 10435057
- [Background] Cheng SP, Liu CL, Liu TP, Hsu YC, Lee JJ. Association between parathyroid hormone levels and inflammatory markers among US adults. Mediators Inflamm. 2014;2014:709024. doi: 10.1155/2014/709024. Epub 2014 Mar 23. PMID 24782595
- [Background] Almqvist EG, Bondeson AG, Bondeson L, Svensson J. Increased markers of inflammation and endothelial dysfunction in patients with mild primary hyperparathyroidism. Scand J Clin Lab Invest. 2011 Apr;71(2):139-44. doi: 10.3109/00365513.2010.543694. Epub 2010 Dec 20. PMID 21166606
- [Background] Emam AA, Mousa SG, Ahmed KY, Al-Azab AA. Inflammatory biomarkers in patients with asymptomatic primary hyperparathyroidism. Med Princ Pract. 2012;21(3):249-53. doi: 10.1159/000334588. Epub 2011 Dec 16. PMID 22179481
- [Background] Rolighed L, Amstrup AK, Jakobsen NF, Sikjaer T, Mosekilde L, Christiansen P, Rejnmark L. Muscle function is impaired in patients with "asymptomatic" primary hyperparathyroidism. World J Surg. 2014 Mar;38(3):549-57. doi: 10.1007/s00268-013-2273-5. PMID 24101026